CLINICAL TRIAL: NCT06007937
Title: A Phase 1/2 Study of Combination Lorlatinib and Ramucirumab in Patients With Advanced ALK-rearranged Lung Cancers
Brief Title: A Study of Lorlatinib in Combination With Ramucirumab in People With Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-131
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer; Metastatic; Recurrent
Keywords: Lorlatinib; Ramucirumab; 23-131
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Recurrence | interventions — lorlatinib; Ramucirumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lorlatinib and ramucirumab (Experimental): The phase 1 safety portion of the study will assess whether a dose of lorlatinib 100 mg orally daily and ramucirumab 10 mg/kg intravenous infusion once every three weeks is a tolerable and safe dose. Six patients will be enrolled at this dose level and assessed for dose limiting toxicities (DLTs) for one full cycle (21 days). Once the phase 1 portion of the study is complete, patients will be enrolled in the phase 2 portion of the study, cohort expansion at the MTD. Patients will be enrolled in two patient cohorts: cohort 1, treatment-naïve and cohort 2, patients who have progressed on prior second-generation ALK TKI. A cycle will be 21 days in length. Response to therapy will initially be assessed by interval imaging every 2 cycles.
  Interventions: Drug: Lorlatinib; Drug: Ramucirumab

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib 100 mg orally daily
Drug: Ramucirumab — Ramucirumab 10 mg/kg intravenous infusion once every three weeks is a tolerable and safe dose.

SUMMARY:
This study will test the safety of the combination of ramucirumab and lorlatinib. The researchers will test one or two different doses of lorlatinib in combination with ramucirumab to find the drug combination dose that causes few or mild side effects in participants. Once the researchers find this dose, they can test it in future participants to see if it is effective in treating their metastatic ALK-rearranged NSCLC. The researchers are also looking to see whether there are specific genes or DNA sequences associated with a response to treatment with lorlatinib and ramucirumab.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >18 years old
* Metastatic or recurrent, biopsy-proven non-small cell lung cancer
* ALK fusion identified by next generation sequencing (NGS) or IHC on material obtained from tumor or plasma
* Measurable (RECIST 1.1) indicator lesion not previously irradiated
* Karnofsky performance status (KPS) ≥ 70%
* Adequate organ function defined as follows: ANC ≥1.5 × 10^9 /L, platelets ≥100 × 10^9/L, hemoglobin ≥ 9 g/dL, INR ≤ 1.5, PTT or aPTT <1.5x ULN, total bilirubin ≤ 1.5 × ULN (Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted), AST ≤ 3 × ULN, ALT ≤ 3 × ULN or ≤ 5 x ULN in the setting of liver metastases, Cr ≤1.5 ULN or CrCl ≥ 40 mL/min. If Cr is

  ≥ 1.5x ULN, a 24-hr urine collection to calculate creatinine clearance must be performed

  °The patient's urinary protein is ≤1+ on dipstick or routine urinalysis (UA); if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol).
* Patients on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight heparin for a minimum of 14 days prior to trial enrollment without signs of active bleeding or pathological condition that carries a high risk of bleeding (eg, tumor invading major vessels or known varices). Patients on warfarin must have an INR ≤ 3.0
* Patients must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] version 5 Grade ≤1) from the acute effects of prior therapy, except for residual alopecia or peripheral neuropathy (up to grade 2 allowed)prior to start of therapy
* Patients in cohort 1 will be treatment-naïve in the metastatic setting. Prior treatment with adjuvant chemotherapy is allowed
* Patients in cohort 2 will have progressed or be intolerant of at least one second generation ALK TKI, including alectinib, brigatinib, or ceritinib.
* Patients may have received multiple ALK TKIs as well as chemotherapy, but one of these treatments must have been with a second-generation ALK TKI.
* Because the teratogenicity of ramucirumab is not known, the patient, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods).
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to first dose of protocol therapy.

Exclusion Criteria:

* Prior lorlatinib or ramucirumab exposure
* Symptomatic, unstable brain metastasis requiring therapy with steroids or radiation therapy. Patients with clinically stable brain metastases (previously treated or untreated) are eligible
* Women who are breastfeeding or pregnant
* Major radiotherapy within 2 weeks of starting treatment on protocol
* Major surgery within 4 weeks of starting treatment on protocol or minor surgery/subcutaneous venous access device placement within 7 days prior to the first dose of protocol therapy
* Less than 3 weeks since previous chemotherapy, 4 weeks since immunotherapy, and 2 weeks from any investigational therapy
* Significant bleeding disorders or grade ≥3 bleeding episode within 12 weeks prior to enrollment. Patients with history of gross hemoptysis (defined as bright red blood of ≥1/2 teaspoon) within 8 weeks prior to enrollment will be excluded
* New or history of diagnosis of deep vein thrombosis (DVT) or pulmonary embolism (PE) or other significant thromboembolic event in the 12 weeks prior to first dose of protocol therapy. Patients with thromboembolic events diagnosed >12 weeks prior to protocol therapy are eligible if on stable doses of anticoagulation as outlined above. Venous port or catheter thrombosis or superficial venous thrombosis are not considered significant events
* GI perforation and/or fistula or bowel obstruction within 6 months or risk factors for perforation prior to enrollment
* Child-Pugh B or greater cirrhosis or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Uncontrolled hypertension, defined as systolic BP ≥160 mm Hg or diastolic BP ≥100 mm Hg, prior to initiating study treatment, despite hypertensive intervention
* Serious or non-healing wound, ulcer or bone fracture within 28 days of enrollment
* Radiologically documented evidence of major blood vessel invasion or encasement by cancer or radiographic evidence of intratumor cavitation
* Active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* Arterial thrombotic event or arterial thromboembolic event, including myocardial infarction, unstable angina, congestive heart failure ≥ NYHA class III, cerebrovascular accident or transient ischemic attack, within 6 months prior to enrollment
* Planned elective or major surgery during the trial
* Chronic therapy with any of the following within 7 days of enrollment:

  * Antiplatelet agents (such as clopidogrel, ticlopidine, dipyridamole, or anagrelide)
  * Aspirin up to 325 mg/day is permitted
* Serious uncontrolled medical disorders or psychological conditions that would, in the opinion of the investigator, limit the patient's ability to complete the study or sign an informed consent document
* Patients with unavoidable strong CYP3A inducer or inhibitor use (see table 15.4 for list of agents)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2028-08-17 (Estimated); Study Completion 2028-08-17 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase I) | 1 year
  Dose limiting toxicities using the NCI Common Terminology Criteria for Adverse Events Version 5 (NCI-CTCAE) will be used to grade toxicities during the trial.
Progression-free survival (Phase II) | 12 months
  by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Riely, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering West Harrison (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm